CLINICAL TRIAL: NCT01760863
Title: The Utility of Oral Antibiotic Therapy Following 2-stage Revision Arthroplasty for Infected Prosthetic Hips and Knees
Brief Title: Oral Antibiotics After 2-Stage Revision for Infected Total Hip Arthroplasty and Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Craig J Della Valle, MD, MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11040802
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Prosthesis-Related Infections
Keywords: Revision; Knee; Hip; Arthroplasty; Oral; Antibiotics; Infection
MeSH Terms: conditions — Prosthesis-Related Infections; Infections | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Antibiotics (Experimental): Oral antibiotics for 3 months; recommendation for antibiotics will be made by an infectious disease specialist.
  Interventions: Other: Oral Antibiotics
- No oral antibiotics (No Intervention): No oral antibiotics.

INTERVENTIONS:
Other: Oral Antibiotics — Oral Antibiotics will be prescribed for 3 months per recommendations of an infectious disease specialist.
  Arms: Oral Antibiotics

SUMMARY:
The primary purpose of this study is to compare the re-infection rates in patients undergoing 2-stage revision arthroplasty who receive additional oral antibiotic therapy to those patients who received in-hospital perioperative antibiotic only. Patients will be monitored for re-infection following hospital discharge, defined as deep infection of the joint space/capsule that requires return to the operating room within 24-months of the re-implantation procedure.

ELIGIBILITY:
Inclusion criteria:

Adult patients undergoing 2-stage revision arthroplasty of the knee or hip with the causative organism(s) identified using tissue culture and/or joint fluid analysis that is amenable to oral antibiotic therapy. Patients must be able to tolerate oral antibiotics and agree to participate in the study.

Exclusion criteria:

Patients with a fungal prosthetic joint infection, unable to tolerate or refuse to undergo oral antibiotic therapy, unable to follow-up at the specified intervals, allergic to the therapy of preference, or have an organism that is not amenable to oral antibiotic therapy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Infection Rate | 24 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Rush University Medical Center, Chicago, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - Rothman Institute, Philadelphia, Pennsylvania
  - Vanderbilt, Nashville, Tennessee

REFERENCES:
- [Result] Zywiel MG, Johnson AJ, Stroh DA, Martin J, Marker DR, Mont MA. Prophylactic oral antibiotics reduce reinfection rates following two-stage revision total knee arthroplasty. Int Orthop. 2011 Jan;35(1):37-42. doi: 10.1007/s00264-010-0992-x. Epub 2010 Mar 7. PMID 20213514